CLINICAL TRIAL: NCT02683811
Title: A Randomised Controlled Study for Evaluating the Effectiveness of the Updated Version of Diario Della Salute, a School-based Program for Prevention of Unhealthy and Risky Behaviours and Promotion of Well-being in Italian Pre-adolescents
Brief Title: Effectiveness of the Updated Version of the School-based Program Diario Della Salute (DDS-2)
Acronym: DDS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale CN2 Alba-Bra (Other)
Collaborators: Eclectica Sas di Beccaria Franca, Ermacora Antonella e C. (Industry); University of Turin, Italy (Other); University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Laura Marinaro, Dr Laura Marinaro, Azienda Sanitaria Locale CN2 Alba-Bra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASLCN2
Record Dates: First submitted 2015-12-18; First posted 2016-02-17 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Adolescent Behavior; Health Behavior; Mental Health Wellness 1
Keywords: adolescence; prevention; wellbeing; evaluation; effectiveness; school-based program
MeSH Terms: conditions — Adolescent Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Diario della Salute (DDS-2), a school-based program aimed to promote psychological well-being and to prevent cigarette smoking, alcohol abuse, unhealthy eating habits, physical inactivity in preadolescents aged 11-13 years. The program is composed by 5 highly standardised interactive units led by previously trained teachers during school hours (15 hours total). Units focus on emotional and social issues related to adolescent developmental tasks. The goal is to promote the adolescent emotional and social skills.
  Interventions: Behavioral: Diario della Salute (DDS-2)
- Control group (No Intervention): No intervention aimed at preventing cigarette smoking, alcohol abuse, unhealthy eating habits, physical inactivity and promoting emotional and social well-being is administered at school by teachers.

INTERVENTIONS:
Behavioral: Diario della Salute (DDS-2) — The updated version of Diario della Salute program (DDS-2) includes: 1) teachers' manual, 2) a booklet for teens telling the story of four same-age students (e.g. experimenting with risky behaviours, conflicting feelings and thoughts, need for independence and control, etc.), 3) a booklet for parents telling the experience of a mum and a dad with teenage children (e.g. problems in the relationship with teenage children, family conflicts, parental control and supervision, family communication, etc.).
  Other Names: Percorsi di promozione del benessere tra i pre-adolescenti
  Arms: Intervention group

SUMMARY:
This study evaluates the short- and long-term effects on psychological wellbeing and health-related behaviours of the updated version of a universal school-based program called Diario della Salute (DDS-2) in Italian students aged 11-13 years.

DETAILED DESCRIPTION:
The updated version of Diario della Salute (DDS-2) is a universal school-based intervention aimed at promoting psychological and emotional well-being and preventing unhealthy and risky behaviours (cigarettes smoking, alcohol abuse, unhealthy eating habits, physical inactivity) in preadolescence. The program is composed by 5 highly standardized interactive units delivered by previously trained teachers during school hours on emotional and social issues related to developmental tasks in adolescence. The kit includes: 1) a teacher's manual, 2) a booklet for each participating student, 3) a booklet for parents of each participating student. The objective is to promote and reinforce adolescents' emotional and social skills as factors contributing to adolescent well-being and health.

A randomised controlled trial with two parallel groups is performed, with 1:1 allocation ratio, in two different Regions of Italy (Piedmont and Veneto). Schools are randomly assigned to one of the two groups (DDS-2 intervention vs. no intervention) and are used as the unit of allocation. Individual participants (i.e. students) are the unit of analysis. Schools are matched by number of students and average socioeconomic status. Eligible schools are identified from the list of all schools having students from 11 to 13 located in study sites. A number of eligible schools accounting for the requested number of students in the target grades is invited to participate in the study. If a school does not respond to the invitation or declines to participate, the school recruitment process is repeated, and another eligible school is invited to participate. The process continues until achievement of the sample size. No incentive is offered to students, families and schools for participating in the study.

A paper-and-pencil self-report anonymous questionnaire developed by the research group is used to determine whether the interventions have changed the outcomes. The questionnaire will be administered in classes by the researchers at baseline, at the end of the intervention and one-year after the end of the intervention (at equal intervals both in the intervention and in the control group). The questionnaire consists of the following sections: 1) demographics, 2) emotional and social skills, 3) psychological wellbeing, 4) school experience, 5) unhealthy and risky behaviours, 6) prosocial and aggressive behaviours. Questionnaires are linked through an anonymous self-generated code.

ELIGIBILITY:
Inclusion Criteria:

1. public/government schools,
2. at least two classes attended by students aged 11-13,
3. not participating in other school-based programs with similar objectives targeted to the classes of interest,
4. providing consensus to study participation. In participating schools, all classes of students aged between 11 and 13 years are eligible to be enrolled in the study.

Exclusion Criteria:

1. private schools,
2. less than two classes attended by students aged 11-13,
3. involved in other school-based programs with similar objectives targeted to the classes of interest. In participating schools, students whose parents opt out from the study are excluded.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3600 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Psychological well-being (Brief Psychological Wellbeing Inventory) | one month after intervention completion
  Four scales (3 items per scale) from Brief Psychological Wellbeing Inventory (PWB, Ryff & Keyes, 1995 - Italian version by Cicognani, Zani, 1999) assessing different areas of perceived wellbeing such as autonomy, environmental mastery, positive relations with others, self-acceptance
Psychosomatic disorders (Health Behaviors in School-aged Children - Symptom checklist) | one month after intervention completion
  8 items from the Italian version of HBSC (Health Behaviors in School-aged Children - Symptom checklist (Haugland et al., 2001; Raves-Sieberer et al., 2009) assessing the frequency of perceived psychological and somatic disorders
Health status (Health Behaviors in School-aged Children Questionnaire) | one month after intervention completion
  1 item from the Italian version of HBSC (Health Behaviors in School-aged Children) Questionnaire assessing the general perceived health status.

SECONDARY OUTCOMES:
Verbal and physical aggression (Verbal and Physical Aggression Scale) | one month after intervention completion
  20 items from Verbal and Physical Aggression Scale (Caprara & Pastorelli, 1988) assessing the frequency of aggressive behaviors
Prosocial behaviours (Prosocial Behaviours Scale) | one month after intervention completion
  15 item from Prosocial Behaviours Scale (Caprara & Pastorelli, 1988) assessing the frequency of prosocial behaviours
School success (Health Behavior Questionnaire) | one month after intervention completion
  1 item from the Health Behavior Questionnaire (Jessor et al., 1992 - Italian version by Bonino et al., 2003) assessing the school performance
Cigarette smoking (HBSC Questionnaire) | one month after intervention completion
  3 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing cigarette smoking behavior
Frequency of cigarette smoking (HBSC Questionnaire) | one month after intervention completion
  1 item from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the number of smoked cigarettes in the last month
Alcohol use (HBSC Questionnaire) | one month after intervention completion
  3 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the use of alcohol
Drunkenness (HBSC Questionnaire) | one month after intervention completion
  3 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the frequency of drunkenness
Eating habits (HBSC Questionnaire) | one month after intervention completion
  16 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the frequency of use of healthy and unhealthy food
Eating style (HBSC Questionnaire) | one month after intervention completion
  2 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the frequency of healthy and unhealthy eating habits per week
Physical activity (HBSC Questionnaire) | one month after intervention completion
  4 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the frequency of physical activity per week
Physical inactivity (HBSC Questionnaire) | one month after intervention completion
  6 items from the Italian version of HBSC (Health Behaviours in School-aged Children) Questionnaire assessing the frequency of sedentary behaviours per day

OTHER OUTCOMES:
Emotional skills (Self- Efficacy Scale) | one month after intervention completion
  27 items from the Italian version of Self- Efficacy Scale (Bandura, 1997 - Italian version by Caprara et al., 2001) assessing the perceived individual emotional skills
Satisfaction with school (School Situation Questionnaire) | one month after intervention completion
  4 scales (5 items per scale) from the School Situation Questionnaire (Santinello & Bertarelli, 2002) assessing the quality of relationship with schoolmates and teachers, self-esteem at school, attitude towards learning
Social skills (Self- Efficacy Scale) | one month after intervention completion
  13 27 items from the Italian version of Self- Efficacy Scale (Bandura, 1997 - Italian version by Caprara et al., 2001) assessing the perceived individual social skills

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marinaro, Principal Investigator — ASL CN2
Locations (5):
- Italy (5):
  - ASL AL, Casale Monferrato, AL
  - Azienda Sanitaria Locale CN2 Alba-Bra, Alba, Cuneo
  - ASL CN1, Cuneo, Cuneo
  - ASL TO1, Torino, Torino
  - Regione Veneto, Venezia, Venezia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: project web site — http://www.diariodellasalute.it/
- Available data/document: Study Protocol — http://www.diariodellasalute.it — Study protocol (Italian version) can be requested by contacting the project manager (lmarinaro@aslcn2.it)
- Available data/document: program materials and tools — http://www.diariodellasalute.it — The Italian version of program materials and tools (teachers' manual, students' booklet and parents' booklet) can be freely accessed and downloaded from project web site.